CLINICAL TRIAL: NCT06410352
Title: Effectiveness of Pharmacologic, Surgical, and Dietetic Weight Loss Methods on Lifespan in Patients With Metabolic Syndrome: a Comparative Clinical Trial
Brief Title: Effectiveness of Weight Loss Methods on Lifespan for Metabolic Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center, Kazakhstan (Other)
Collaborators: Nazarbayev University School of Medicine (Unknown); Nazarbayev University (Other); Astana Medical University (Other); Public Association "Eurasian Society of Personalized Medicine" (Unknown); Ministry of Science and Higher Education of the Republic of Kazakhstan (Other Government)
Responsible Party: Principal Investigator, Kuat Oshakbayev, full-Professor, University Medical Center, Kazakhstan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP23488544
Record Dates: First submitted 2024-04-29; First posted 2024-05-13 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; obesity; type 2 diabetes mellitus; weight loss; telomere length; quality of life; cost effectiveness analysis
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Diabetes Mellitus, Type 2; Weight Loss | interventions — semaglutide; empagliflozin

STUDY DESIGN:
Intervention Model Description: One of the methods that will be used in project is a new drug combination for weight loss in patients with T2D - Glucagon-like-peptide-1-receptor-agonists with sodium-glucose-co-transporter-2-inhibitors. Guidelines on hyperglycemic management recommend either GLP-1RAs or SGLT-2is as second-line treatments for patients with T2D on metformin monotherapy. The use of both antidiabetic drugs in combination is rare in the literature. During the last decade, the results of large-scale, randomized, clinical trials on newer antidiabetic agents, GLP-1RA and SGLT-2 inhibitor have been shown to modify cardiovascular risk factors, such as insulin resistance, body weight, BP, and lipid profile, additionally to induce weight loss.
  The second method is a bariatric operation - minigastric bypass (MGB) that is endovideososcopic techniques with the intraperitoneal using of synthetic/biological materials. MGB is performed to reduce the absorption surface of the gastrointestinal
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pharmacologic weight loss (Combination Product) (Active Comparator): The 1st group (n=50) receives subcutaneous Semaglutide (GLP-1RA) 1 mg once a 7 day with oral Empagliflozin (SGLT-2i) 25 mg once a day that is a novel combination additionally to standard medical treatment including anti-diabetes, antihypertensive, lipid-lowering, symptomatic therapy.
  Interventions: Drug: Semaglutide, Empagliflozin
- Surgical weight loss (Active Comparator): The 2nd group (n=50) receives surgical method (laparoscopic MGB). These patients pass through additional pre-operation examination (blood tests and electrocardiography, esophagogastroscopy, ultrasound, and other necessary standard methods).
  Interventions: Procedure: Minigastric bypass
- Very-low-calorie-restriction diet (Experimental): The 3rd group (n=50) receives very-low-calorie-restriction diet ('Analimentary-detoxication') including <100 kcal/day with fat-free vegetables (tomato/cucumber) and salt intake (5-6 g/day), optimum physical activity, and sexual self-restraint. The program goals the next outputs: a) use of own fatty store; b) control endogen intoxication; c) reuse of interim metabolic substrates.
  Interventions: Dietary Supplement: Analimentary detoxication
- Ramadan fast's weight loss (Experimental): The 4th group (n=30) adheres to fasting on Ramadan fast (RF) season. They strictly adhered to two principles of nutrition during RF: 1) "no blood, no smell of fat" which means "don't eat meat and don't eat fatty foods"; 2) the 'Sehri time' (a meal eaten before dawn) included just 1.5-2.0 glass of water and fruits of 80-100 gr (apple, dates, and persimmon). Indeed, the patients followed a diet in which they ate one meal a day - participants have a meal during 'Iftar time' (a meal eaten after sunset).
  Interventions: Behavioral: Ramadan fast's weight loss

INTERVENTIONS:
Drug: Semaglutide, Empagliflozin — subcutaneous Semaglutide (GLP-1RA) 1 mg once a 7 day with oral Empagliflozin (SGLT-2i) 25 mg once a day
  Other Names: Semaglutide (GLP-1RA), Empagliflozin (SGLT-2i)
  Arms: Pharmacologic weight loss (Combination Product)
Procedure: Minigastric bypass — Endovideososcopic techniques with the intraperitoneal using of synthetic/biological materials. MGB is performed to reduce the absorption surface of the gastrointestinal tract by shunting the greater part of the stomach, the duodenum and the initial section of the small intestine, which reduces the absorption of food and leads to a decrease in the production of gastrointestinal hormones.
  Other Names: bariatric operation
  Arms: Surgical weight loss
Dietary Supplement: Analimentary detoxication — very-low-calorie-restriction diet ('Analimentary-detoxication') including <100 kcal/day with fat-free vegetables (tomato/cucumber) and salt intake (5-6 g/day), optimum physical activity, and sexual self-restraint.
  Other Names: Very-low-calorie diet
  Arms: Very-low-calorie-restriction diet
Behavioral: Ramadan fast's weight loss — The participants adhered to fasting on RF season. They strictly adhered to two principles of nutrition during RF: 1) "no blood, no smell of fat" which means "don't eat meat and don't eat fatty foods"; 2) the 'Sehri time' (a meal eaten before dawn) included just 1.5-2.0 glass of water and fruits of 80-100 gr (apple, dates, and persimmon). Indeed, the patients followed a diet in which they ate one meal a day - participants have a meal during 'Iftar time' (a meal eaten after sunset).
  Other Names: Ramadan fast
  Arms: Ramadan fast's weight loss

SUMMARY:
Background. The prevalence of type 2 diabetes mellitus (T2D) in the world is constantly increasing. Treatment of T2D is complicated by arterial hypertension and obesity (metabolic syndrome - MS). Cardiovascular complications are the main cause of death in patients with MS. Objective weight loss improves clinical and laboratory parameters in patients with T2D and hypertension.

Purpose: To study lifespan, glycemic and lipid metabolism, quality of life, and cost-effectiveness of pharmacologic, surgical, and dietetic weight loss methods in obese patients with MS at 24 weeks in a comparative clinical trial.

Methods:

1. st stage - Study design: An open pilot prospective clinical trial. The study included 71 adult patients with T2D and hypertension for the Ramadan fast's (RF) weight loss.
2. nd stage - Study design: A 24-week open label, prospective, multicenter, comparative clinical trial with the intention-to-treat analysis.

Participants. Totally 150 adult patients with MS aged 35-65 years and with BMI≥27 kg/m2 for Asian will be included. They will be distributed in three comparative groups: drug treatment, surgery and diet.

Primary endpoints: weight loss, fasting blood glucose, blood insulin level, systolic/diastolic BP.

Secondary endpoints: blood lipids, heel bone mineral density (HBMD), and ejection fraction (EF).

Expected results:

A prospective multicenter clinical study will provide comparative results on life expectancy, glycemic and lipid metabolism, quality of life, cost-effectiveness of pharmacological, bariatric and dietary methods of weight loss in patients with obesity, T2D and hypertension. As a result of the research, the following will be published:

1. at least three articles and/or reviews in peer-reviewed scientific publications indexed in the Science Citation Index Expanded of the Web Of Science database and/or having a Cite Score percentile in the Scopus of at least 50;
2. at least 1 patent for an invention (including a positive decision on it).

DETAILED DESCRIPTION:
At the 1 st stage of the study will screen 71 adult patients for eligibility aged 35 to 65 years with T2D and hypertension for the RF. T2D was treated with Metformin, Sulfonylurea, GLP-1 agonists (exenatide, liraglutide), Glitazones in different combinations; hypertension was treated with beta-blockers, calcium channel blockers, diuretics, SGLT-2 Inhibitors (empagliflozin, canagliflozin) in different combinations. Patients with heart failure (HF) in their medical records and anamnesis with reduced ejection fraction <55% also will be included; I-II stages of the NYHA functional classification.

Inclusion criteria: 1) written informed consent; 2) 35≤ age <65 years old; 2) any BMI and WC; 3) diagnosis of T2D and hypertension ≥3 years and treatment with non-hormonal conventional pharmacological medications; 4) any level of triglycerides, cholesterol, body fat%; 5) weight loss on the RF for 30 days.

Exclusion criteria: 1) age <35 or ≥65 years old; 1) Insulin-depended T2D and uncontrolled high BP; 2) patients taking gastrointestinal lipase inhibitors, etc.; 3) presence of acute infection diseases or exacerbation of chronic diseases; 4) ejection fraction <30%; 5) history of alcohol consumption >30 g/day within the past 5 years; 6) malignancy within the past 5 years; gestation or lactation; kidney failure; hereditary diseases; or known hypersensitivity to any of the test substances.

Outcome measures: Primary endpoints: weight loss, fasting blood glucose, blood insulin level, systolic/diastolic BP. Secondary endpoints: blood lipids, heel bone mineral density (HBMD), and EF.

Intervention. The participants adhered to fasting on RF season. They strictly adhered to two principles of nutrition during RF: 1) "no blood, no smell of fat" which means "don't eat meat and don't eat fatty foods"; 2) the 'Sehri time' (a meal eaten before dawn) included just 1.5-2.0 glass of water and fruits of 80-100 gr (apple, dates, and persimmon). Indeed, the patients followed a diet in which they ate one meal a day - participants have a meal during 'Iftar time' (a meal eaten after sunset). The participants also adhered to walking at least 3,000 steps/day, sexual self-restraint.

A combination of in-person conversations and telephone calls conductes during the 30-day study period: the baseline/7-day/14-day and 30-day RF.

At the 2nd stage of the study will include totally 150 adult patients with MS distributed in three comparative groups: drug treatment, surgery and diet therapy.

The study design is prospective because the investigators have to comparatively measure TL before/after interventions; the study may not be an observation study. Because of the trial will non-randomized patients will be allocated to each group based on equal baseline characteristics according to the inclusion/exclusion criteria and including adjustments for baseline and confounding characteristics.

The patients will be allocated to each group based on the patient and two physicians (surgeon and therapist) decisions to avoid the risk of "selection bias". Normalization of parameters will focuse on the work required to embed processes into statistics.

Inclusion criteria: 1) written informed consent; 2) T2D≥3-year with glucose lowering therapy including insulin; 3) 35-55 years old; 4) BMI≥27 kg/m2 for both sex, for Asian ethnicity; 5) ongoing treatment with antihypertensive treatment; 6) weight loss 15-20% at baseline and dynamic follow-up up to 24 weeks.

All included patients before recruiting to the study received standard-of-care treatment for T2D and AH according to regional guidelines.

Exclusion criteria: T1D; <34 age >56 years old; unstable cardiac disorders (New York Heart Association class IV heart failure, refractory angina, uncontrolled arrhythmias, critical valvular heart disease, or severe uncontrolled hypertension); glomerular filtration rate <30 mL/min and/or dialysis within 14 days before screening; malignancy within the past 5 years; gestation or lactation; hereditary diseases; known hypersensitivity to any of the test substances.

The 1st group (n=50) receives subcutaneous Semaglutide (GLP-1RA) 1 mg once a 7 day with oral Empagliflozin (SGLT-2i) 25 mg once a day that is a novel combination additionally to standard medical treatment including anti-diabetes, antihypertensive, lipid-lowering, symptomatic therapy.

The 2nd group (n=50) receives surgical method (laparoscopic MGB). These patients pass through additional pre-operation examination (blood tests and electrocardiography, esophagogastroscopy, ultrasound, and other necessary standard methods).

The 3rd group (n=50) receives very-low-calorie-restriction diet ('Analimentary-detoxication') including <100 kcal/day with fat-free vegetables (tomato/cucumber) and salt intake (5-6 g/day), optimum physical activity, and sexual self-restraint. The program goals the next outputs: a) use of own fatty store; b) control endogen intoxication; c) reuse of interim metabolic substrates.

A combination of in-person conversations and telephone calls conduct during the study period.

Justification of the sample size. The estimated treatment difference will set to 10% with a standard deviation of 8% and the superiority margin of 5% (δ=0.05) based on two-sided hypothesis testing. Using SPSS,Sample-Power,V23.0, the number of evaluable individuals needed per treatment arm >32. At least 150 patients will be screened and recruited in the comparative clinical trial.

End Points: The primary endpoints: reduction in body weight 15-20% from baseline; leukocyte TL. The secondary endpoints: HbA1c; fasting blood glucose and 2-hour oral glucose tolerance test (OGTT); systolic/diastolic BP; lipid profile; immunoassay insulin in blood; adverse events.

Methods:

* Criteria for the diagnosis of MS. Diagnosis of MS (IDF-2005). Diagnosis T2D: HbA1c≥6,5%, fasting plasma glucose level ≥7.0 mmol/l, or a patient receives antidiabetic therapy [ADA, 2023]. [55] AH: systolic-BP≥130 and/or their diastolic-BP≥90 mm.Hg following repeated examination, or a patient receives antihypertensive-drugs.
* General obesity will be measured by determining of BMI (kg/m2). Abdominal obesity is assessed by waist circumference using the standards for the Asian nationality by IDF(2018). [56]
* Body composition parameters including fat mass, visceral fat, fat-free mass, total body-water, muscle/bone mass, metabolic age, basal-metabolic-rate, and bioimpedance will be evaluated by Tanita-MC-980MA Multi-Frequency Segmental Body-Composition-Analyzerer(TanitaCorp,Japan).
* Physical activity will be assessed as the number of steps taken by patients, as determined by individual pedometers from Hoffmann-La-Roche(Switzerland) or other individual digital system.
* Laboratory study. On the same blood samples, standard laboratory a complete blood count, erythrocyte sedimentation rate, urea, creatinine, glucose, electrolytes, HbA1c, lipid profile (total-cholesterol, HDL/LDL, triglycerides), total proteins, coagulation profile, bilirubin, hepatic enzyme activities, blood/ urine ketone bodies.
* Hormones assay. Fasting serum insulin by immunoassay method (CzechRepublic). The Homeostasis Model Assessment insulin resistance indexes (HOMA-IR) will be used as a surrogate measure of insulin sensitivity as follows: HOMA-IR=((fasting insulin in nU/L)×(fasting glucose in mmol/l)/22.5).
* Measurement of TL. TL will be measured in T/S ratio with an adaptation of the quantitative polymerase chain reaction (q-PCR) methods. The intraassay and interassay variability (CV) for quantitative polymerase chain reaction will be shown.

Blood samples for measurement of TL will be collected in sterile vacutainer and delivered to the Genom and personalized medicine laboratory (Nazarbayev University). DNA was purified using Promega Wisard DNA system in -20 С. In short, for measurement of telomere repeat copies, primers will be added. Two control samples will be run in each experiment to allow for normalization between experiments, and periodical reproducibility experiments will be performed to guarantee correct measurements. The ratio calculated is proportional to average TL per cell.

* Quality of life assesses with international questionnaire BAROS Bariatric Analysis and Reporting Outcome System, EuroQoL.
* Cost-effectiveness analysis conductes using as outcomes both clinical as well as EuroQol to estimate the incremental cost-effectiveness of the three alternative interventions. Analysis considers specific costs (a) direct medical costs (including the intervention itself and follow-up care to the condition), (b) indirect nonmedical costs, and (c) additional non-medical costs. Costs of medical care obtaines from economic departments of participating medical centers identifying resources consumed during the interventions. Indirect costs obtaines from patients. The limited time horizon of this study will make it necessary to use a model to extrapolate the observed effect of the treatments assessed in the long term.
* Consultations of specialists conductes before/during/after the study 24-week period.
* Imaging methods: Ultrasound of internal organs (GE Vivid 7 Ultrasound; GE Healthcare Worldwide USA, Michigan); ECG.

Interpretation of the data. The primary hypothesis is that patients treated with the comparative methods would experience a greater weight reduction and improving in the primary/secondary endpoints; then the groups selects to compare between themselves in the aggregate using multiple linear regression analysis. To establish the effectiveness of the comparative methods based on the principle: H0 (null hypothesis) one method doesn't differ from another/other; and Ha (alternative) one method differs from another/other.

Statistical analysis. The statistical analysis plan considers non-compliance, loss-of-follow-up, and missing-data. Multiple-logistic-regression-models, ANOVA/ANCOVA uses to predict the probability of specific variables. Mixed-effect-models or generalized-estimating-equations (GEE) evaluates with statisticians. The Student's two-factor-t-test, OR (95%,CI), Pearson's criterion-χ2 will be used to assess differences in proportions. Mann-Whitney U-test and Kruskal-Wallis test are used for nonparametric. Pearson or Spearman correlation coefficient (r). To determine dependent/independent variables and to control confounders discusses between the team using literature data.

Regression analysis performs using state of the art machine learning algorithms in python code. These include application of algorithms such as KNN, SVM and Random Forests. Additionally, the investigators will apply deep learning methodology for creating a model to test the hypothesis testing as a binary classifier. This learning model uses neural network, given new data will be able to make personalized effects of the three treatment methods. Study data presentes in tables as M±SE or median (25-75%) based on distribution of variables. Survival analysis (Kaplan-Meier or Cox-regression) uses to assess mortality in the three comparative treatments. Statistical analysis using SPSS for Windows,ver.28.0.

Ethics. The appropriate national and institutional regulatory authorities and ethics committees will approve the study design, and all participants will provide written informed consent. The study will fulfilled in University Medical Center together with Nazarbayev University School of Medicine and National Laboratory Astana and Astana Medical University.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent;
* T2D≥3-year with glucose lowering therapy including insulin;
* 35-55 years old;
* BMI≥27 kg/m2 for both sex, for Asian ethnicity;
* ongoing treatment with antihypertensive treatment;
* weight loss 15-20% at baseline and dynamic follow-up up to 24 weeks.

Exclusion Criteria:

* T1D;
* <34 age >56 years old;
* unstable cardiac disorders (New York Heart Association class IV heart failure, refractory angina, uncontrolled arrhythmias, critical valvular heart disease, or severe uncontrolled hypertension);
* glomerular filtration rate <30 mL/min and/or dialysis within 14 days before screening; • malignancy within the past 5 years;
* gestation or lactation;
* hereditary diseases;
* known hypersensitivity to any of the test substances.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Weight | Baseline, 24 weeks
  weight in kilograms
Body mass index | Baseline, 24 weeks
  weight and height will be combined to report BMI in kg/m^2
Fat mass | Baseline, 24 weeks
  fat mass in % of total body weight and total kg
Fat free mass | Baseline, 24 weeks
  fat free mass in % of total body weight and total kg
blood insulin level | Baseline, 24 weeks
  Fasting serum insulin (nU/L) was determined by immunoassay (Immunotech Insulin Irma kit, Prague, Czech Republic)
systolic/diastolic Blood presure | Baseline, 24 weeks
  Blood pressure is measured in units of millimeters of mercury (mmHg). The readings are always given in pairs, with the upper (systolic) value first, followed by the lower (diastolic) value.
Fasting blood glucose | Baseline, 24 weeks
  mmol per liter

SECONDARY OUTCOMES:
Total cholesterol | Baseline, 24 weeks
  Total cholesterol in mmol/l
HbA1c | Baseline, 24 weeks
  glycosilated hemoglobin in % or/and mmol/mol
Triglycerides | Baseline, 24 weeks
  Triglycerides in gr/L
High-density lipoprotein | Baseline, 24 weeks
  high-density lipoprotein i n mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Kuat Oshakbayev, professor, Principal Investigator — University Medical Center, Kazakhstan
Locations (1):
- Kuat Pernekulovich Oshakbayev, Astana, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No
The de-personalized data will be available from the authors upon reasonable request. Those wishing to request the study data should contact Principal Investigator of a research grant: Dr. Oshakbayev Kuat